CLINICAL TRIAL: NCT05240274
Title: A Single Site, Placebo Controlled, Double Blind Randomised Clinical Trial Evaluating the Effectiveness of Metformin to Prevent Post-transplant Diabetes in a Cohort of Patients Undergoing Renal Transplantation
Brief Title: The POWERED Study: Prophylaxis With Metformin to Prevent PTDM
Acronym: POWERED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 203080
Record Dates: First submitted 2022-01-17; First posted 2022-02-15 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-11

CONDITIONS: Post-transplant Diabetes Mellitus; New Onset Diabetes After Transplant; New Onset Diabetes After Transplantation; Kidney Transplant; Complications; Renal Transplantation; End Stage Renal Disease; Metformin
Keywords: post-transplant diabetes mellitus; new onset diabetes after transplant; renal transplant; kidney transplant; end-stage kidney disease; metformin; PTDM; NODAT
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Single site, placebo controlled, double blind randomised clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the patient and the study team will be blinded to the treatment intervention. The clinical team will also be blinded.
  Pharmacy staff who dispense the IMP will not be blinded, nor will Sponsor Office staff responsible for reporting unblinded SUSAR reports to the MHRA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): metformin 500mg OD
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): placebo 500mg OD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — metformin 500mg OD for 3 months to start within 10 days post-renal transplant
  Arms: Metformin
Drug: Placebo — placebo 500mg OD for 3 months to start within 10 days post-renal transplant
  Arms: Placebo

SUMMARY:
PrOphylaxis With mEtformin to pREvent PTDM: a single site, placebo controlled, double blind randomised clinical trial evaluating the effectiveness of metformin to prevent post-transplant diabetes in a cohort of patients undergoing renal transplantation.

DETAILED DESCRIPTION:
Renal transplantation is the optimal form of renal-replacement therapy in end-stage kidney disease. However, up to 30% of new renal transplants develop post-transplant diabetes mellitus (PTDM). The development of PTDM is associated with adverse graft and patient survival outcomes and represents an increased financial burden. There is an urgent clinical need to discover therapies which could decrease the risk of developing PTDM. Metformin offers a safe and cheap therapeutic option which has been demonstrated to reduce the incidence of type 2 diabetes in a high-risk non-transplant patient group. The investigators propose to study its safety and efficacy in preventing the development of PTDM.

POWERED is a single site, placebo-controlled, double- blind randomised clinical trial of metformin in patients without pre-existing diabetes mellitus who have received a new renal transplant. Eligible, consented patients are randomised to a 3 month course of either active drug or placebo within 10 days post-transplant. All patients will receive the usual standard of care for transplant patients. Clinical and laboratory data will be collected and assessed at baseline and throughout their participation in the study. The primary endpoint is the development of PTDM as defined by a positive oral glucose tolerance test (OGTT). Secondary endpoints include graft outcomes, pancreatic b-cell function and safety endpoints. The study began recruitment in January 2019 and plans to enrol 60 patients. There are no interim analyses planned.

Ethical approval was obtained from the London - Brighton and Sussex Ethics Committee (REC 18/LO/0958) prior to commencing the study. All study-related data will be used by the Sponsor in accordance with local data protection law. Results of the trial will be submitted for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) undergoing renal transplantation under the care of the Barts Health NHS Trust Renal Department
2. Aged 18-75 inclusively
3. Willing to comply with study schedule

Exclusion Criteria:

1. History of Type 1 or type 2 diabetes
2. Clinically significant history of abnormal physical and/or mental health as judged by the investigator other than conditions related to chronic kidney disease
3. Participation in an investigational drug trial in the 3 months prior to administration of the initial dose of study drug
4. Subject with a known hypersensitivity or contraindication to Tacrolimus
5. Subject with a known hypersensitivity or contraindication to Metformin
6. Pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis of post-transplant diabetes | 12 months post-renal transplant
  Positive 2 hour oral glucose tolerance test (i.e. 2 hour sugar >11.1 mol/L)

SECONDARY OUTCOMES:
Pancreatic beta cell function | 12 months
  change in calculated HOMA-IR using C-peptide measurement between baseline and month 3 using
HbA1c | 12 months
  HbA1c
impaired glucose tolerance | 12 months
  impaired glucose tolerance as per 2 hour oral glucose tolerance test (i.e. 2 hour glucose 7.9-11.1 mmol/L)
patient and graft survival | 12 months
  patient survival, kidney transplant (graft) survival
incidence of treatment emergent adverse events | 12 months
  patient safety: adverse events, serious adverse events
rejection | 12 months
  episodes of acute transplant rejection
eGFR | 12 months
  renal transplant function
diagnosis of PTDM in OGTT screen fails | 12 months
  incidence of PTDM in patients not randomised to study due to positive OGTT at screening: defined by appearance of PTDM on problem list or prescription of an anti-diabetic drug

CONTACTS AND LOCATIONS:
Overall Officials: Kieran McCafferty, M.B., B.Chir, Principal Investigator — Barts Health NHS Trust; Queen Mary University London
Locations (1):
- Royal London Hospital, Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any published article, after de-identification (text, tables, figures, and appendices).
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  The data may be used for individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found by emailing the corresponding author.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT05240274/Prot_SAP_000.pdf